CLINICAL TRIAL: NCT01610661
Title: Dietary Carbohydrate Type and CVD Risk Indicators
Brief Title: Dietary Carbohydrate Type and Cardiovascular Disease (CVD) Risk Indicators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2735
Record Dates: First submitted 2011-11-07; First posted 2012-06-04 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Dyslipidemia
Keywords: carbohydrate; inflammation; glucose homeostasis; gene expression
MeSH Terms: conditions — Dyslipidemias; Inflammation | interventions — Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Unrefined-carbohydrate (Other): unrefined carbohydrate diet
  Interventions: Other: Diet
- Refined-carbohydrate (Other): refined carbohydrate diet
  Interventions: Other: Diet
- Simple-carbohydrate (Other): simple carbohydrate diet
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Unrefined-carbohydrate refers to foods made with 100% whole grains (wheat, rice, corn). Refined-carbohydrate refers to foods made with white flour (e.g., bread, pasta) or white rice. Simple-carbohydrate refers to foods made with sucrose (50% glucose/50% fructose) and high-fructose corn syrup.
  Other Names: simple carb; refined carb; unrefined carb

SUMMARY:
The aim of this study is to determine the effect of habituation to diets with different types of carbohydrate (simple-carb, refined-carb, unrefined-carb) on selected Cardiovascular Disease (CVD) risk indicators.

DETAILED DESCRIPTION:
The objective of this pilot study is to determine the relative comparability for an isocaloric exchange of (1) refined-carb for simple-carb and (2) refined-carb for unrefined-carb, on established and emerging CVD risk indicators. To achieve this goal, subjects with moderate dyslipidemia (LDL cholesterol > 100mg/dL) will consume diets enriched in 3 types of carbohydrate (simple-carb, refined-carb and unrefined-carb) according to a randomized, cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* LDL cholesterol (>100 mg/dL)
* > 50 years (all females postmenopausal, as defined by complete natural cessation of menses for > 12 months or a bilateral oophorectomy)
* BMI > 25 and < 35 kg/m2
* Normal kidney function as assessed by serum creatinine and blood urea nitrogen
* Normal liver function as assessed by serum glutamic oxaloacetic transaminase and alkaline phosphatase
* Normal thyroid function as assessed by serum thyroid stimulating hormone concentrations
* Normal gastrointestinal function
* Fasting plasma glucose concentrations < 120 mg/dL
* Normotensive with or without medication
* Non-smoker for at least 12 months
* Alcohol intake of less than 7 drinks per week
* Consistent physical activity pattern

Exclusion Criteria:

* < 50 years old
* BMI < 25 and > 35 kg/m2
* LDL cholesterol <100 mg/dL
* Abnormal fasting plasma glucose levels >120 mg/dL
* Use of medications known to affect lipid metabolism:

  * Bile Acid Sequestrants (Cholestyramine, Colestipol, Colesevelam, etc.)
  * Cholesterol Absorption Inhibitors (Ezetimibe [Zetia])
  * Nicotinic Acid Agents (Niacin, Niacor, Slo-Niacin, etc)
  * Fibrates (Gemfibrozil [Lopid], Ciprofibrate, Fenofibrate [Tricor], etc)
  * Probucol
* Use of anticoagulants (Coumadin, Heparin, Plavix, etc), anabolic steroids, and hydrocortisone
* Use of hormone therapy medications containing estrogen
* Use of fish oil / omega-3 supplements, and Metamucil (or fiber containing dietary supplements)
* Any Aspirin, non-steroidal anti-inflammatory drugs (NSAID) or antihistamine use or therapies that cannot be discontinued by subject for 72 hours prior to blood draws and adipose tissue collection and any NSAIDS for 72 hours after the procedure for obtaining adipose tissue sample
* Established cardiovascular disease as defined by history of myocardial infarction, stroke, heart failure, coronary artery bypass graft, stenosis >50%, angina and peripheral arterial disease
* Uncontrolled hypertension or high blood pressure reading at the discretion of the study physician or nurse
* Renal or kidney disease, as defined by a history of chronic kidney disease or by glomerular filtration rate of < 60 ml.min/1.73 m2 calculated from screening blood tests
* Liver disease, as defined by a history of chronic hepatitis B or C, cholestatic or cirrhotic liver disease, nonalcoholic fatty liver disease, elevations of serum glutamic-pyruvic transaminase (SGPT) or serum glutamic oxaloacetic transaminase (SGOT) greater than 1.5 times the upper limit of normal at screening, bilirubin greater than 2 mg/dL (in the absence of benign causes of elevated bilirubin such as Gilbert's syndrome) at screening, or albumin below the lower limit of normal
* Hypothyroidism or hyperthyroidism, defined as screening TSH outside of normal ranges (<0.4 or >4.5), unless controlled with medication for at least 6 months
* Type I and II diabetes
* Gastrointestinal disease
* Lidocaine Allergy
* Smoking within the past 12 months.
* Alcohol intake > 7 drinks per week or unwillingness to not consume alcohol while participating in the study
* Unwillingness to maintain body weight during participation in the study
* Unwillingness to adhere to diet and study protocol
* Weight gain or loss of more than 15 lb within 6 months prior to enrollment
* Non-English speaking subjects
* No Social Security number
* Food allergies or aversions
* Blood donation within the past 8 weeks

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-04 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
fasting plasma lipid profile | 15-week period

SECONDARY OUTCOMES:
glucose | 15 week period
insulin | 15-week period
adipose tissue inflammatory markers | 15-week period
gut microbiome | 15-week period
High-sensitivity C-reactive protein(hsCRP) | 15-week period
Interleukin 6 (IL-6) | 15-week period
Monocyte Chemoattractant Protein 1 (MCP-1) | 15-week period
Tumor necrosis factor-alpha (TNF-alpha) | 15-week period
Monocyte gene expression | 15-week period

CONTACTS AND LOCATIONS:
Overall Officials: Alice H. Lichtenstein, D.Sc., Principal Investigator — Tufts University
Locations (1):
- Jean Mayer Human Nutrition Research Center on Aging, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Faits T, Walker ME, Rodriguez-Morato J, Meng H, Gervis JE, Galluccio JM, Lichtenstein AH, Johnson WE, Matthan NR. Exploring changes in the human gut microbiota and microbial-derived metabolites in response to diets enriched in simple, refined, or unrefined carbohydrate-containing foods: a post hoc analysis of a randomized clinical trial. Am J Clin Nutr. 2020 Dec 10;112(6):1631-1641. doi: 10.1093/ajcn/nqaa254. PMID 32936872
- [Derived] Meng H, Matthan NR, Fried SK, Berciano S, Walker ME, Galluccio JM, Lichtenstein AH. Effect of Dietary Carbohydrate Type on Serum Cardiometabolic Risk Indicators and Adipose Tissue Inflammatory Markers. J Clin Endocrinol Metab. 2018 Sep 1;103(9):3430-3438. doi: 10.1210/jc.2018-00667. PMID 29982704